CLINICAL TRIAL: NCT02017483
Title: Explore the Association Between the Emotion Recognition and the Attention Processing Under the Emotional Stimuli in ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201211008RIB
Record Dates: First submitted 2013-12-04; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: ADHD,; emotion recognition; attention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Lots of studies suggest that children with ADHD have deficits in facial emotion recognition, especially for the negative emotion. But there were arguments for this deficit is a secondary problem due to the general attention impairment in ADHD, or a specific social cognitive processing to ADHD. The objectives of this study are to investigate that association between the deficits in facial emotion recognition and the emotional attention processing in ADHD. In this study, the investigators use the emotion attentional bias and emotional go / no go paradigm to answer this question.

DETAILED DESCRIPTION:
The sample will consist of 100 children and adolescent with ADHD and 100 typical controls, ages 8-16. The ADHD group inclusion criteria are patients who have clinically diagnosis of DSM-IV ADHD confirmed by the K-SADS-E, and have IQ > 80; and whose parents consent to this study.

The measurements will be included:

1. Diagnostic assessment tools:

   * Chinese version of Kiddie-Schedule for Affective Disorders and Schizophrenia-Epidemiology version.
   * Conners' Parent/Teacher Rating Scale- Revised: Short Form, CPRS-R:S/CTRS-R:S.
   * Swanson, Nolan, and Pelham, Version Ⅳ（SNAP-Ⅳ）Rating Scale - Parent/ Teacher Form.
2. Emotion assessment tools:

   * Facial emotion recognition task.
   * Emotional attentional bias task.
   * Emotional Go/ No Go task.
3. Cognitive assessment tool:

   * Wechsler Intelligence Scale for Children-Fourth Edition Chinese Version.

This study could offer the suggestion for the further intervention of social function in ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Control group

   * The subjects without ADHD.
   * Ages range from 8 to 16
   * Full scale IQ ≥ 80
   * The subjects who and whose parents consent to this study.
2. ADHD group

   * Patients who have clinically diagnosis of DSM-IV ADHD confirmed by the K-SADS-E.
   * Ages range from 8 to 16
   * Full scale IQ ≥ 80
   * Patients who and whose parents consent to this study.

Exclusion Criteria:

* Mental Retardation
* Schizophrenia, Schizoaffective Disorder
* Mood Disorders
* Organic Psychosis
* Learning Disorder
* Pervasive Developmental Disorder
* The subjects of control group if have a history of the following condition as defined by DSM-IV: ADHD in addition to the above exclusion criteria will be excluded.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will recruit 100 children and adolescent with ADHD and 100 typical controls.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The error rate in facial emotion judgements on computerized task | up to 2 years
  Investigator used the e-prime program to assess the error rate in facial emotion judgements. Participants need to judge the emotion of the face stimuli presented on the laptop.

SECONDARY OUTCOMES:
The reaction time of attentional bias for pairs of face stimuli(happy/neutral or angry/neutral faces) on dot-prob task | up to 2 years
  Investigator presented pairs of face stimuli with emotional and neutral expressions and probed the allocation of attention to these stimuli for presentation times of 150 and 500 ms to assess the reaction time of attentional bias. Participants need to press the dot after the prob.

OTHER OUTCOMES:
The attentional inhibition control(omission errors and commission errors) in emotional go/no go task | up to 2 years
  Investigator used go/ no go task to assess participants' omission errors and commission errors, participants just need to press the keyboard and the number of errors were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan